CLINICAL TRIAL: NCT03333291
Title: Characterisations of Microbial Community Composition and Kinetics Following Faecal Microbiota Transplantation in Patients WITH IRRITABLE BOWEL SYNDROME
Brief Title: Fecal Transplantation in Patients With IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Vest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/1497
Record Dates: First submitted 2017-10-25; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Open pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fecal transplantation (Experimental): Duodenal transfer of healthy donor fecal suspension
  Interventions: Dietary Supplement: fecal suspension

INTERVENTIONS:
Dietary Supplement: fecal suspension — helathy donor fecal suspension administered by duodenal scope

SUMMARY:
The study will characterize the biology of FMT in the context of IBS prior to wider clinical application of the method. Given the ethical concerns of unknown and long-term adverse effects of FMT therapy, the study will include patients only with moderate to severe symptoms. IBS is a heterogenous disorder and it is important to characterize the patients, and study as homogeneous patient populations as possible. Therefore the study will only include post-infectious IBS patients after the Giardia outbreak.

DETAILED DESCRIPTION:
Primary aims:

Detailed characterisation of donor and recipient microbial community composition (by means of 16S rRNA profiling) and determination of the kinetics of changes following FMT

Secondary aims:

* Determination of interactions of importance to persisting recipient gut microbiota.
* Evaluate safety of FMT in an IBS population
* To evaluate the efficacy of FMT in relieving symptoms in selected patients with IBS in an open pilot trial in order to have the possibility to calculate number of patients needed when planning future controlled studies.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-and 70 years
* IBS-SSS (IBS-Symptom Severity Scale) score >175 (175 - 300 represents moderate, > 300 represent severe IBS).
* All patients are required to have symptoms for at least 12 months, fulfilling the Rome III criteria with either diarrhoea-predominant irritable bowel syndrome (IBS-D) or alternating constipation and diarrhoea (IBS-A) with bloating or flatulence as predominant symptoms. Only IBS considered post-infectious after the Bergen Giardia outbreak will be included. The severity of global IBS symptoms has to be either moderate ("cannot be ignored but do not influence daily activities") or severe ("influence daily activities"). A decrease of 50 points on the IBS-SSS has been shown to correlate with improvement in clinical symptoms. All patients will undergo appropriate investigations to exclude organic disease.

Exclusion Criteria:

* History of inflammatory bowel diseases, gastrointestinal malignancy, blood in stool or antibiotic use within 1 month prior to FMT, immunocompromised patient defined as taking immuno-suppressive medications, history of opportunistic infections within 1 year prior to FMT, oral thrush, or disseminated lymphadenopathy.
* Patients who are scheduled for abdominal surgery, pregnant women or patients taking probiotics or taking antibiotics within 4 weeks prior to installation are also excluded from the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Stool microbiota changes | up to 28 weeks
  abundance of major microbial taxa in fecal transplant post transplantation

SECONDARY OUTCOMES:
Global improvement in IBS symptoms | up to 28 weeks
  Patient questionnaires IBSS-S

CONTACTS AND LOCATIONS:
Locations (1):
- Helse Bergen HF, Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mazzawi T, El-Salhy M, Lied GA, Hausken T. The Effects of Fecal Microbiota Transplantation on the Symptoms and the Duodenal Neurogenin 3, Musashi 1, and Enteroendocrine Cells in Patients With Diarrhea-Predominant Irritable Bowel Syndrome. Front Cell Infect Microbiol. 2021 May 12;11:524851. doi: 10.3389/fcimb.2021.524851. eCollection 2021. PMID 34055657
- [Derived] Mazzawi T, Hausken T, Hov JR, Valeur J, Sangnes DA, El-Salhy M, Gilja OH, Hatlebakk JG, Lied GA. Clinical response to fecal microbiota transplantation in patients with diarrhea-predominant irritable bowel syndrome is associated with normalization of fecal microbiota composition and short-chain fatty acid levels. Scand J Gastroenterol. 2019 Jun;54(6):690-699. doi: 10.1080/00365521.2019.1624815. Epub 2019 Jun 13. PMID 31190584
- [Derived] Mazzawi T, Lied GA, Sangnes DA, El-Salhy M, Hov JR, Gilja OH, Hatlebakk JG, Hausken T. The kinetics of gut microbial community composition in patients with irritable bowel syndrome following fecal microbiota transplantation. PLoS One. 2018 Nov 14;13(11):e0194904. doi: 10.1371/journal.pone.0194904. eCollection 2018. PMID 30427836